CLINICAL TRIAL: NCT04363684
Title: ARTFL LEFFTDS Longitudinal Frontotemporal Lobar Degeneration (ALLFTD)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: University of California, San Francisco (Other); National Institute on Aging (NIA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Bradley Boeve, Principal Investigator, Mayo Clinic
Other Study IDs: 19-004543; U19AG063911 (NIH)
Record Dates: First submitted 2020-04-02; First posted 2020-04-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Frontotemporal Lobar Degeneration (FTLD); Progressive Supranuclear Palsy (PSP); Corticobasal Degeneration (CBD); Behavioral Variant Frontotemporal Dementia (bvFTD); Semantic Variant Primary Progressive Aphasia (svPPA); Nonfluent Variant Primary Progressive Aphasia (nfvPPA); FTD With Amyotrophic Lateral Sclerosis (FTD/ALS); Amyotrophic Lateral Sclerosis; Oligosymptomatic PSP (oPSP); C9orf72; GRN Related Frontotemporal Dementia; MAPT Gene Mutation; TBK1 Gene Mutation; Oligosymptomatic Progressive Supranuclear Palsy
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia With Motor Neuron Disease; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, plasma, serum, PBMC, CSF (CSF is optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Longitudinal Arm: Annual clinic visits throughout the length of the study.
- Biofluid-Focused Arm: Single clinic visit.

SUMMARY:
ARTFL LEFFTDS Longitudinal Frontotemporal Lobar Degeneration (ALLFTD) represents the formalized integration of ARTFL (U54 NS092089; funded through 2019) and LEFFTDS (U01 AG045390; funded through 2019) as a single North American research consortium to study FTLD for 2019 and beyond.

DETAILED DESCRIPTION:
The ARTFL LEFFTDS Longitudinal Frontotemporal Dementia (ALLFTD) study aims to evaluate sporadic (s-) and familial (f-) frontotemporal lobar degeneration (FTLD) patients and asymptomatic family members of f-FTLD patients, characterizing the cohorts longitudinally and informing clinical trial design. The study has two arms: a "longitudinal arm" involving a comprehensive assessment of clinical, functional, imaging, and biofluid data collection annually, and a "biofluid-focused arm" involving limited clinical data to accompany biospecimen collection. For more information: https://www.allftd.org/

ELIGIBILITY:
Longitudinal Arm Inclusion Criteria

Familial FTLD (f-FTLD) participants (either is acceptable):

* members of families in whom at least one member has a known disease-associated mutation in one of the major genes that cause f-FTLD: MAPT, GRN, C9orf72 (or other rare genes)
* an autosomal dominant family history of a FTLD syndrome (without a known gene) verified by medical record review or well-documented family history including family members with a medical history consistent with FTLD or a related disorder.

Sporadic FTLD (s-FTLD) participants:

Sporadic participants should be symptomatic with no known family history nor a genetic mutation indicating f-FTLD. All sporadic participants must have an FTLD syndrome as a referring diagnosis; those determined by ALLFTD clinicians to have non-FTLD diagnoses will be excluded from longitudinal visits, but their baseline visit will be included in comparative datasets. For inclusion in the longitudinal follow-up, participants should meet research criteria for one of the following FTLD syndromes:

* Progressive Supranuclear Palsy (PSP)
* Semantic variant Primary Progressive Aphasia (svPPA)
* Nonfluent variant Primary Progressive Aphasia (nfvPPA)
* Corticobasal Degeneration (CBD)/Corticobasal Syndrome (CBS)
* Behavioral variant Frontotemporal dementia (bvFTD)
* Frontotemporal Dementia with Amyotrophic Lateral Sclerosis (FTD/ALS)

Biofluid-Focused Arm Inclusion Criteria

Participants enrolled in the biofluid arm may be either f-FTLD or s-FTLD. All general inclusion criteria apply. Participants should meet research criteria (as specified above) for any FTLD syndrome or meet familial FTLD inclusion criteria. Because the biofluid arm participants do not undergo the same detailed clinical and functional assessments required for the longitudinal arm, participants may be included regardless of primary language, as long as an appropriately translated consent is available.

Exclusion Criteria:

* Known presence of a structural brain lesion (e.g. tumor, cortical infarct) that could reasonably explain symptoms in a symptomatic participant.
* Known presence of an Alzheimer's disease causing mutation in PSEN1, PSEN2 or APP; or biomarker evidence for Alzheimer's disease as a cause of the clinical syndrome.
* A previous history of Korsakoff encephalopathy, severe alcohol dependence (within 5 years of onset of dementia), frequent alcohol or other substance intoxication, or other neurological disorder.
* Evidence through history or laboratory testing of uncorrected B12 deficiency (B12 < 95% of local laboratory's normal value), unregulated hypothyroidism (TSH >150% of normal), HIV positive, renal failure (creatinine > 2), liver failure (ALT or AST > two times normal), respiratory failure that requires supplemental oxygen, large confluent white matter lesions, significant systemic medical illnesses such as deteriorating cardiovascular disease.
* Current medication likely to affect CNS functions in the opinion of the site PI.
* In the site investigator's opinion, the participant cannot complete sufficient key study procedures. The participant may be enrolled into the biofluid-focused arm if they can tolerate a blood draw and short clinical exam, but must be able to complete at least 75% of study procedures for enrollment into the longitudinal arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will have a referring diagnosis of an FTLD clinical syndrome or will be a member of a family with a strong family history of an FTLD syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Brain Volumes | Baseline, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year
  Compare rates of change in whole brain and regional volumes between asymptomatic f-FTLD and symptomatic f- and s-FTLD, measured using MRI.
Change in NIH Examiner Executive Composite Score | Baseline, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year
  Evaluate change in NIH Examiner Executive Composite Score in asymptomatic f-FTLD.
Change in Multidomain Impairment Rating (MIR) Scale | Baseline, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year
  Annual change in MIR score (total score 0-3), which is a new global scale for FTLD that incorporates behavioral, cognitive, and motor dysfunction in the rating.

SECONDARY OUTCOMES:
Plasma Neurofilament Light Chain Analysis | 5 years
  Annual blood samples will be collected to detect changes in plasma neurofilament light chain concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Boeve, MD, Principal Investigator — Mayo Clinic; Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco; Howie Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (27):
- United States (25):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - NIH, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washinton University in St. Louis, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Nantz National Alzheimer Center Houston, Houston, Texas
  - UT San Antonio Health Science Center, San Antonio, Texas
  - University of Washington, Seattle, Washington
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - University of Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified subject level data will be shared upon approved data request.
Time Frame: De-identified data will be available for at least the duration of the study.
Access Criteria: Interested researchers must complete a data request through the ALLFTD website. All data requests will be reviewed by a committee for evaluation of scientific merit and feasibility. Please consult the website for additional information regarding this process (https://www.allftd.org/policies).
  Approved requests will be delivered in a de-identified manner.
URL: https://www.allftd.org/data

REFERENCES:
- [Derived] Tipton PW, Deutschlaender AB, Savica R, Heckman MG, Brushaber DE, Dickerson BC, Gavrilova RH, Geschwind DH, Ghoshal N, Graff-Radford J, Graff-Radford NR, Grossman M, Hsiung GR, Huey ED, Irwin DJ, Jones DT, Knopman DS, McGinnis SM, Rademakers R, Ramos EM, Forsberg LK, Heuer HW, Onyike C, Tartaglia C, Domoto-Reilly K, Roberson ED, Mendez MF, Litvan I, Appleby BS, Grant I, Kaufer D, Boxer AL, Rosen HJ, Boeve BF, Wszolek ZK; ALLFTD Consortium. Differences in Motor Features of C9orf72, MAPT, or GRN Variant Carriers With Familial Frontotemporal Lobar Degeneration. Neurology. 2022 Sep 13;99(11):e1154-e1167. doi: 10.1212/WNL.0000000000200860. Epub 2022 Jul 5. PMID 35790423
- See also: ALLFTD Study Website — https://www.allftd.org/